CLINICAL TRIAL: NCT00689351
Title: Phase 2, Randomized, Active-Controlled, Double-Blind Trial Evaluating The Safety, Tolerability, And Immunogenicity Of A 13-Valent Pneumococcal Conjugate Vaccine In Healthy Infants Given With Routine Pediatric Vaccinations In Korea
Brief Title: Study Evaluating A 13-Valent Pneumococcal Conjugate Vaccine Administered To Infants In Korea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-010; B1851001
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Pneumococcal Vaccine
Keywords: Prevention; against; pneumococcal; disease; Vaccine
MeSH Terms: conditions — Disease | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 13vPnC
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine
- 2 (Active Comparator): 7vPnC
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — 13vPnC is given via intramuscular injection at approximately 2, 4, 6 and 12 months of age.
  Arms: 1
Biological: 7-valent pneumococcal conjugate vaccine — 7vPnC is given via intramuscular injection at approximately 2, 4, 6 and 12 months of age.
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate vaccine (13vPnC), relative to a 7-valent pneumococcal conjugate vaccine (7vPnC) when given concomitantly with routine vaccines in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2-month-old-infants (42 to 98 days)
* Available for the entire study period (14 months)

Exclusion Criteria:

* Previous vaccine with pneumococcal, diptheria, tetanus, pertussis, polio or Hib vaccine
* A previous severe reaction to any vaccine or vaccine-related component

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- South Korea (6):
  - Pfizer Investigational Site, Incheon, Bupyeong-gu
  - Pfizer Investigational Site, Seoul, Jongno-gu
  - Pfizer Investigational Site, Incheon, Jung-gu
  - Pfizer Investigational Site, Kyunggi, Koyang
  - Pfizer Investigational Site, Seoul, Seodaemun-gu
  - Pfizer Investigational Site, Seoul, Yeongdeungpo-gu

REFERENCES:
- [Derived] Kim DS, Shin SH, Lee HJ, Hong YJ, Lee SY, Choi KM, Oh CE, Kim KH, Juergens C, Patterson S, Giardina PC, Gruber WC, Emini EA, Scott DA. Immunogenicity and safety of 13-valent pneumococcal conjugate vaccine given to korean children receiving routine pediatric vaccines. Pediatr Infect Dis J. 2013 Mar;32(3):266-73. doi: 10.1097/INF.0b013e3182748bb6. PMID 23011012
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-010&StudyName=Study%20Evaluating%20A%2013-Valent%20Pneumococcal%20Conjugate%20Vaccine%20Administered%20To%20Infants%20In%20Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) dose administered intramuscularly (IM) at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose).
Period: Infant Series of Dosing
Arm/Group | 13vPnC | 7vPnC
Started | 91 | 89
Vaccinated Dose 1 | 88 | 89
Vaccinated Dose 2 | 86 | 88
Vaccinated Dose 3 | 85 | 88
Completed | 85 | 88
Not Completed | 6 | 1
Not completed — Parent/legal guardian request | 5 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 85 | 88
Completed | 84 | 88
Not Completed | 1 | 0
Not completed — Parent/legal guardian request | 1 | 0
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 84 | 88
Completed | 84 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 91 | 89 | 180
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.3) | 2.1 (0.2) | 2.1 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 39 | 84
  Male | 46 | 50 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Serotype-specific Immunoglobulin G (IgG) Antibody Level Greater Than or Equal to (≥) 0.35 Micrograms Per Milliliter (Mcg/mL) Measured 1 Month After the Infant Series
Description: Percentage of participants achieving predefined antibody threshold ≥0.35 Mcg/mL along with the corresponding 95 percent (%) confidence interval (CI) was calculated for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A).
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable Infant Immunogenicity population: participants who were 41 to 99 days of age (inclusive) on the day of the first vaccination, who had treatments as randomized (all expected doses) and at least 1 valid and determinate assay result for proposed analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 91 | 89
percentage of participants
  Serotype 4 | 100.0 [95.7 to 100.0] | 100.0 [95.8 to 100.0]
  Serotype 6B | 98.8 [93.5 to 100.0] | 100.0 [95.8 to 100.0]
  Serotype 9V | 100.0 [95.7 to 100.0] | 100.0 [95.8 to 100.0]
  Serotype 14 | 100.0 [95.7 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 18C | 100.0 [95.7 to 100.0] | 100.0 [95.8 to 100.0]
  Serotype 19F | 97.6 [91.6 to 99.7] | 98.8 [93.6 to 100.0]
  Serotype 23F | 98.8 [93.5 to 100.0] | 98.8 [93.6 to 100.0]
  Serotype 1 | 100.0 [95.7 to 100.0] | 2.4 [0.3 to 8.2]
  Serotype 3 | 100.0 [95.7 to 100.0] | 2.4 [0.3 to 8.2]
  Serotype 5 | 100.0 [95.7 to 100.0] | 57.5 [45.9 to 68.5]
  Serotype 6A | 97.6 [91.6 to 99.7] | 72.3 [61.4 to 81.6]
  Serotype 7F | 100.0 [95.7 to 100.0] | 4.8 [1.3 to 11.7]
  Serotype 19A | 100.0 [95.7 to 100.0] | 100.0 [95.6 to 100.0]

2. Secondary Outcome: Percentage of Participants Achieving a Serotype-specific IgG Antibody Level ≥0.35 Mcg/mL Measured 1 Month After the Toddler Dose
Description: Percentage of participants achieving predefined antibody threshold ≥0.35Mcg/mL along with the corresponding 95% CI was calculated for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A). Exact 2-sided CI was based on the observed percentage of participants.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: Evaluable Toddler Immunogenicity population:41-99 days old inclusive on day of first vaccination, 365-395 days old inclusive at toddler dose, had all treatments as randomized, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 91 | 89
percentage of participants
  Serotype 4 | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 6B | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 9V | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 14 | 98.7 [93.1 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 18C | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 19F | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 23F | 100.0 [95.5 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 1 | 100.0 [95.5 to 100.0] | 1.3 [0.0 to 6.9]
  Serotype 3 | 100.0 [95.5 to 100.0] | 12.0 [5.9 to 21.0]
  Serotype 5 | 100.0 [95.5 to 100.0] | 92.4 [84.2 to 97.2]
  Serotype 6A | 98.8 [93.2 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 7F | 100.0 [95.4 to 100.0] | 23.6 [13.2 to 37.0]
  Serotype 19A | 100.0 [95.5 to 100.0] | 98.8 [93.5 to 100.0]

3. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) of Serotype-specific IgG Antibody 1 Month After the Infant Series
Description: Antibody GMC along with corresponding 2-sided 95% CI for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Geometric mean concentrations (GMCs) were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after the infant series (7 months of age)
Population: Evaluable Infant Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 91 | 89
Mcg/mL
  Serotype 4 | 5.40 [4.62 to 6.30] | 6.97 [5.94 to 8.18]
  Serotype 6B | 5.71 [4.64 to 7.03] | 4.88 [3.96 to 6.01]
  Serotype 9V | 3.33 [2.90 to 3.83] | 3.78 [3.31 to 4.33]
  Serotype 14 | 14.83 [12.38 to 17.77] | 16.29 [13.36 to 19.85]
  Serotype 18C | 4.57 [3.98 to 5.24] | 4.73 [4.09 to 5.47]
  Serotype 19F | 3.88 [3.18 to 4.72] | 4.20 [3.55 to 4.96]
  Serotype 23F | 4.29 [3.56 to 5.16] | 4.11 [3.40 to 4.98]
  Serotype 1 | 7.44 [6.25 to 8.85] | 0.02 [0.02 to 0.03]
  Serotype 3 | 1.60 [1.35 to 1.89] | 0.04 [0.03 to 0.05]
  Serotype 5 | 5.06 [4.37 to 5.85] | 0.39 [0.30 to 0.49]
  Serotype 6A | 5.73 [4.64 to 7.07] | 0.64 [0.49 to 0.82]
  Serotype 7F | 6.97 [6.07 to 8.00] | 0.04 [0.03 to 0.05]
  Serotype 19A | 5.94 [5.13 to 6.89] | 2.65 [2.29 to 3.06]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Serotype 4: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.77, 95% CI 2-sided [0.62 to 0.97] — CI for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC, 7vPnC)
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Serotype 6B: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 1.17, 95% CI 2-sided [0.87 to 1.57] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Serotype 9V: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.88, 95% CI 2-sided [0.73 to 1.07] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Serotype 14: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.91, 95% CI 2-sided [0.70 to 1.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Serotype 18C: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.97, 95% CI 2-sided [0.79 to 1.18] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Serotype 19F: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.92, 95% CI 2-sided [0.71 to 1.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Serotype 23F: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 1.04, 95% CI 2-sided [0.80 to 1.36] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Serotype 1: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 329.44, 95% CI 2-sided [242.98 to 446.67] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Serotype 3: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 40.79, 95% CI 2-sided [30.27 to 54.97] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Serotype 5: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 13.12, 95% CI 2-sided [9.92 to 17.34] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Serotype 6A: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 9.01, 95% CI 2-sided [6.46 to 12.56] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; Serotype 7F: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 165.90, 95% CI 2-sided [122.95 to 223.85] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; Serotype 19A: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 2.24, 95% CI 2-sided [1.83 to 2.75] — [estimate comment as in outcome 3, analysis 1]

4. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) of Serotype-specific IgG Antibody 1 Month After the Toddler Dose
Description: as for outcome 3
Time Frame: 1 month after the Toddler Dose (13 months of age)
Population: Evaluable Toddler Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 91 | 89
Mcg/mL
  Serotype 4 | 6.46 [5.29 to 7.90] | 8.25 [6.88 to 9.89]
  Serotype 6B | 16.81 [14.36 to 19.68] | 15.14 [11.91 to 19.25]
  Serotype 9V | 4.59 [3.91 to 5.38] | 4.83 [4.12 to 5.67]
  Serotype 14 | 11.51 [9.59 to 13.80] | 15.64 [13.07 to 18.72]
  Serotype 18C | 6.86 [5.67 to 8.29] | 7.44 [6.27 to 8.83]
  Serotype 19F | 7.75 [6.30 to 9.53] | 5.35 [4.52 to 6.33]
  Serotype 23F | 10.95 [8.77 to 13.66] | 10.44 [8.60 to 12.68]
  Serotype 1 | 9.29 [7.65 to 11.28] | 0.04 [0.03 to 0.05]
  Serotype 3 | 1.65 [1.40 to 1.95] | 0.10 [0.08 to 0.13]
  Serotype 5 | 8.92 [7.62 to 10.45] | 1.31 [1.09 to 1.56]
  Serotype 6A | 13.58 [11.28 to 16.36] | 3.33 [2.67 to 4.14]
  Serotype 7F | 11.17 [9.33 to 13.37] | 0.10 [0.07 to 0.14]
  Serotype 19A | 10.12 [8.55 to 11.98] | 2.38 [2.04 to 2.78]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Serotype 4: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.78, 95% CI 2-sided [0.60 to 1.02] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Serotype 6B: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 1.11, 95% CI 2-sided [0.83 to 1.48] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Serotype 9V: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.95, 95% CI 2-sided [0.76 to 1.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Serotype 14: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.74, 95% CI 2-sided [0.57 to 0.95] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Serotype 18C: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 0.92, 95% CI 2-sided [0.72 to 1.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Serotype 19F: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 1.45, 95% CI 2-sided [1.11 to 1.88] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Serotype 23F: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 1.05, 95% CI 2-sided [0.78 to 1.40] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Serotype 1: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 234.33, 95% CI 2-sided [176.33 to 311.41] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Serotype 3: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 16.63, 95% CI 2-sided [12.19 to 22.69] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Serotype 5: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 6.84, 95% CI 2-sided [5.39 to 8.67] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Serotype 6A: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 4.08, 95% CI 2-sided [3.07 to 5.43] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; Serotype 7F: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 110.92, 95% CI 2-sided [77.09 to 159.59] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC vs 7vPnC; Serotype 19A: Ratio of geometric means (13vPnC, 7vPnC); Test type: Superiority or Other; Student t distribution; Geometric mean ratio computed using Student t distribution for the mean difference of the measures on the log scale; Ratio of geometric means = 4.25, 95% CI 2-sided [3.39 to 5.33] — [estimate comment as in outcome 3, analysis 1]

5. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 1 (2 Months of Age)
Description: Pre-specified local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (greater than [>] 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 1 (2 months of age)
Population: Safety population: All participants who received at least 1 dose of the study vaccine; N=number of participants reporting yes for at least 1 day or no for all days; n=number of participants reporting the specific characteristic.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 75 | 79
percentage of participants
  Tenderness: Any (n=23,26) | 31.9 | 34.2
  Tenderness: Significant (n=6,2) | 8.8 | 2.8
  Swelling: Any (n=14,18) | 19.7 | 24.7
  Swelling: Mild (n=8,18) | 11.6 | 24.7
  Swelling: Moderate (n=7,4) | 10.1 | 5.7
  Redness: Any (n=27,22) | 37.5 | 29.3
  Redness: Mild (n=23,19) | 32.9 | 25.3
  Redness: Moderate (n=4,3) | 5.8 | 4.3
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any tenderness; Test type: Superiority or Other; p = 0.862, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for significant tenderness; Test type: Superiority or Other; p = 0.157, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any swelling; Test type: Superiority or Other; p = 0.550, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild swelling; Test type: Superiority or Other; p = 0.052, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate swelling; Test type: Superiority or Other; p = 0.366, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any redness; Test type: Superiority or Other; p = 0.301, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild redness; Test type: Superiority or Other; p = 0.362, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate redness; Test type: Superiority or Other; p = 0.718, Fisher Exact

6. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 2 (4 Months of Age)
Description: Pre-specified local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 cm to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 2 (4 months of age)
Population: Safety; N=number of participants reporting yes for at least 1 day or no for all days; n=number of participants reporting the specific characteristic.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 62 | 68
percentage of participants
  Tenderness: Any (n=23,24) | 38.3 | 37.5
  Tenderness: Significant (n=0,3) | 0.0 | 5.0
  Swelling: Any (n=22,18) | 35.5 | 28.6
  Swelling: Mild (n=18,15) | 29.5 | 24.6
  Swelling: Moderate (n=4,4) | 7.1 | 6.6
  Redness: Any (n=20,25) | 32.8 | 38.5
  Redness: Mild (n=18,24) | 29.5 | 36.9
  Redness: Moderate (n=4,3) | 7.1 | 5.1
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any tenderness; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for significant tenderness; Test type: Superiority or Other; p = 0.245, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any swelling; Test type: Superiority or Other; p = 0.447, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild swelling; Test type: Superiority or Other; p = 0.684, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate swelling; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any redness; Test type: Superiority or Other; p = 0.578, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild redness; Test type: Superiority or Other; p = 0.451, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate redness; Test type: Superiority or Other; p = 0.712, Fisher Exact

7. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 6
Time Frame: Within 4 days after dose 3 (6 months of age)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 66 | 64
percentage of participants
  Tenderness: Any (n=15,16) | 23.4 | 27.1
  Tenderness: Significant (n=0,1) | 0.0 | 1.9
  Swelling: Any (n=18,14) | 27.7 | 23.3
  Swelling: Mild (n=13,13) | 21.0 | 22.0
  Swelling: Moderate (n=7,4) | 11.3 | 7.0
  Redness: Any (n=19,16) | 30.2 | 26.2
  Redness: Mild (n=12,15) | 20.0 | 25.0
  Redness: Moderate (n=7,3) | 11.5 | 5.6
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any tenderness; Test type: Superiority or Other; p = 0.681, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for significant tenderness; Test type: Superiority or Other; p = 0.482, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any swelling; Test type: Superiority or Other; p = 0.683, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild swelling; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate swelling; Test type: Superiority or Other; p = 0.533, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any redness; Test type: Superiority or Other; p = 0.692, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild redness; Test type: Superiority or Other; p = 0.662, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate redness; Test type: Superiority or Other; p = 0.331, Fisher Exact

8. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Toddler Dose (12 Months of Age)
Description: as for outcome 6
Time Frame: Within 4 days after toddler dose (12 months of age)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 57 | 57
percentage of participants
  Tenderness: Any (n=19,14) | 33.9 | 25.9
  Tenderness: Significant (n=3,1) | 5.9 | 2.0
  Swelling: Any (n=11,10) | 22.4 | 18.9
  Swelling: Mild (n=4,7) | 8.2 | 13.5
  Swelling: Moderate (n=9,4) | 18.4 | 7.8
  Swelling: Severe (n=1,0) | 2.0 | 0.0
  Redness: Any (n=15,12) | 28.8 | 22.2
  Redness: Mild (n=9,10) | 17.6 | 18.5
  Redness: Moderate (n=8,3) | 16.0 | 6.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any tenderness; Test type: Superiority or Other; p = 0.409, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for significant tenderness; Test type: Superiority or Other; p = 0.617, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any swelling; Test type: Superiority or Other; p = 0.807, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild swelling; Test type: Superiority or Other; p = 0.527, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate swelling; Test type: Superiority or Other; p = 0.144, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for severe swelling; Test type: Superiority or Other; p = 0.495, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for any redness; Test type: Superiority or Other; p = 0.506, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for mild redness; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for moderate redness; Test type: Superiority or Other; p = 0.200, Fisher Exact

9. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Infant Series Dose 1 (2 Months of Age)
Description: Pre-specified systemic events (any fever ≥ 38 degrees Celsius [C], decreased appetite, irritability, increased sleep, and decreased sleep) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 4 days after dose 1 (2 months of age)
Population: Safety; N=number of participants reporting yes for at least 1 day or no for all days; n=number of participants reporting the event.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 83 | 86
percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C (n=11,9) | 15.9 | 12.5
  Decreased appetite (n=23,22) | 32.4 | 28.9
  Irritability (n=38,56) | 49.4 | 70.9
  Increased sleep (n=37,30) | 49.3 | 39.0
  Decreased sleep (n=28,38) | 37.8 | 50.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for fever ≥38 degrees C but but less than or equal to (≤)39 degrees C; Test type: Superiority or Other; p = 0.633, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased appetite; Test type: Superiority or Other; p = 0.721, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for irritability; Test type: Superiority or Other; p = 0.009, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for increased sleep; Test type: Superiority or Other; p = 0.253, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased sleep; Test type: Superiority or Other; p = 0.143, Fisher Exact

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Infant Series Dose 2 (4 Months of Age)
Description: as for outcome 9
Time Frame: Within 4 days after dose 2 (4 months of age)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 64 | 72
percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C (n=6,8) | 10.9 | 13.1
  Decreased appetite (n=16,28) | 27.1 | 44.4
  Irritability (n=25,36) | 40.3 | 53.7
  Increased sleep (n=17,16) | 28.8 | 26.2
  Decreased sleep (n=18,27) | 30.0 | 40.9
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for fever ≥38 degrees C but ≤39 degrees C; Test type: Superiority or Other; p = 0.781, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased appetite; Test type: Superiority or Other; p = 0.060, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for irritability; Test type: Superiority or Other; p = 0.159, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for increased sleep; Test type: Superiority or Other; p = 0.839, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased sleep; Test type: Superiority or Other; p = 0.264, Fisher Exact

11. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Infant Series Dose 3 (6 Months of Age)
Description: as for outcome 9
Time Frame: Within 4 days after dose 3 (6 months of age)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 65 | 64
percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C (n=8,5) | 13.6 | 9.3
  Fever >39 degrees C but ≤40 degrees C (n=0,1) | 0.0 | 2.0
  Decreased appetite (n=14,16) | 23.0 | 28.1
  Irritability (n=13,25) | 21.0 | 41.7
  Increased sleep (n=18,12) | 29.5 | 21.1
  Decreased sleep (n=10,17) | 16.4 | 29.3
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for fever ≥38 degrees C but ≤39 degrees C; Test type: Superiority or Other; p = 0.563, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for fever >39 degrees C but ≤40 degrees C; Test type: Superiority or Other; p = 0.468, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased appetite; Test type: Superiority or Other; p = 0.535, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for irritability; Test type: Superiority or Other; p = 0.019, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for increased sleep; Test type: Superiority or Other; p = 0.398, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased sleep; Test type: Superiority or Other; p = 0.125, Fisher Exact

12. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events: Toddler Dose (12 Months of Age)
Description: as for outcome 9
Time Frame: Within 4 days after toddler dose (12 months of age)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 64 | 65
percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C (n=7,10) | 13.7 | 19.6
  Fever >39 degrees C but ≤40 degrees C (n=1,0) | 2.0 | 0.0
  Decreased appetite (n=13,15) | 22.8 | 27.8
  Irritability (n=18,21) | 30.5 | 37.5
  Increased sleep (n=11,8) | 21.2 | 15.4
  Decreased sleep (n=11,20) | 20.4 | 34.5
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for fever ≥38 degrees C but ≤39 degrees C; Test type: Superiority or Other; p = 0.596, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for fever >39 degrees C but ≤40 degrees C; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased appetite; Test type: Superiority or Other; p = 0.663, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for irritability; Test type: Superiority or Other; p = 0.439, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for increased sleep; Test type: Superiority or Other; p = 0.613, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Comparison between treatments for decreased sleep; Test type: Superiority or Other; p = 0.138, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline through 1 Month after last study vaccination (13 Months). Local reactions and systemic events assessed within 4 days of dose: Infant Series Dose 1=2 months of age; Dose 2=4 months of age; Dose 3=6 months of age; Toddler Dose=12 months of age.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Groups:
- Infant Series 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) dose administered intramuscularly (IM) at 2, 4, and 6 months of age (infant series).
- Infant Series 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series).
- After the Infant Series 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series); assessment 1 month after the infant series (7 months of age).
- After the Infant Series 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered IM at 2, 4, and 6 months of age (infant series); assessment 1 month after the infant series (7 months of age).
- Toddler Dose 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5mL dose administered IM at 12 months of age (toddler dose).
- Toddler Dose 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC ) 0.5mL dose administered IM at 12 months of age (toddler dose).
Arm/Group | Infant Series 13vPnC | Infant Series 7vPnC | After the Infant Series 13vPnC | After the Infant Series 7vPnC | Toddler Dose 13vPnC | Toddler Dose 7vPnC
Serious Adverse Events (participants affected / at risk) | 8/88 | 9/89 | 9/88 | 12/89 | 3/84 | 3/88
Other Adverse Events (participants affected / at risk) | 78/88 | 75/89 | 18/88 | 19/89 | 28/84 | 36/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (N=88) | Infant Series 7vPnC (N=89) | After the Infant Series 13vPnC (N=88) | After the Infant Series 7vPnC (N=89) | Toddler Dose 13vPnC (N=84) | Toddler Dose 7vPnC (N=88)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 2 | 4 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 1 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 3 | 2 | 1 | 0
Kawasaki's disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0
Herpangina (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infant Series 13vPnC (N=88) | Infant Series 7vPnC (N=89) | After the Infant Series 13vPnC (N=88) | After the Infant Series 7vPnC (N=89) | Toddler Dose 13vPnC (N=84) | Toddler Dose 7vPnC (N=88)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 4 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 4 | 2 | 0 | 0 | 1 | 0
Dacryostenosis acquired (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Entropion (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 10 | 3 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 8 | 4 | 0 | 1 | 3 | 2
Injection site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atopy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 24 | 30 | 3 | 4 | 7 | 10
Bronchiolitis (Infections and infestations) | 17 | 9 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 11 | 17 | 3 | 0 | 3 | 9
Bronchitis (Infections and infestations) | 10 | 10 | 2 | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 12 | 7 | 0 | 0 | 4 | 2
Otitis media acute (Infections and infestations) | 9 | 5 | 0 | 1 | 0 | 4
Pharyngotonsillitis (Infections and infestations) | 4 | 1 | 1 | 1 | 1 | 3
Acute tonsillitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpangina (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Periorbital cellulit (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Perineal fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 | 16 | 1 | 2 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 17 | 2 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Grunting (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 | 8 | 2 | 4 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 7 | 3 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 6 | 2 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tenderness (any) (Skin and subcutaneous tissue disorders) | 23/72 | 26/76 | 0/0 | 0/0 | 19/56 | 14/54 — Infant Series Dose 1 and Toddler Dose; tenderness (any)=present at site of vaccination
Tenderness (any) (Skin and subcutaneous tissue disorders) | 23/60 | 24/64 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; tenderness (any)=present at site of vaccination
Tenderness (any) (Skin and subcutaneous tissue disorders) | 15/64 | 16/59 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; tenderness (any)=present at site of vaccination
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 6/68 | 2/72 | 0/0 | 0/0 | 3/51 | 1/50 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 0/55 | 3/60 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)=present and interfered with limb movement
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 0/58 | 1/54 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)=present and interfered with limb movement
Swelling (any) (Skin and subcutaneous tissue disorders) | 14/71 | 18/73 | 0/0 | 0/0 | 11/49 | 10/53 — Infant Series Dose 1 and Toddler Dose; Swelling (any)=present at site of vaccination
Swelling (any) (Skin and subcutaneous tissue disorders) | 22/62 | 18/63 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (any)=present at site of vaccination
Swelling (any) (Skin and subcutaneous tissue disorders) | 18/65 | 14/60 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (any)=present at site of vaccination
Swelling (mild) (Skin and subcutaneous tissue disorders) | 8/69 | 18/73 | 0/0 | 0/0 | 4/49 | 7/52 — Infant Series Dose 1 and Toddler Dose; Swelling (mild)=0.5 to 2.0 cm
Swelling (mild) (Skin and subcutaneous tissue disorders) | 18/61 | 15/61 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (mild)=0.5 to 2.0 cm
Swelling (mild) (Skin and subcutaneous tissue disorders) | 13/62 | 13/59 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (mild)=0.5 to 2.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 7/69 | 4/70 | 0/0 | 0/0 | 9/49 | 4/51 — Infant Series Dose 1 and Toddler Dose; Swelling (moderate)=2.5 to 7.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 4/56 | 4/61 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (moderate)=2.5 to 7.0 cm
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 7/62 | 4/57 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (moderate)=2.5 to 7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/67 | 0/70 | 0/0 | 0/0 | 1/49 | 0/50 — Infant Series Dose 1 and Toddler Dose; Swelling (severe) >7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/55 | 0/59 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Swelling (severe) >7.0 cm
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/58 | 0/53 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Swelling (severe) >7.0 cm
Redness (any) (Skin and subcutaneous tissue disorders) | 27/72 | 22/75 | 0/0 | 0/0 | 15/52 | 12/54 — Infant Series Dose 1 and Toddler Dose; Redness (any)=present at site of vaccination.
Redness (any) (Skin and subcutaneous tissue disorders) | 20/61 | 25/65 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (any)=present at site of vaccination
Redness (any) (Skin and subcutaneous tissue disorders) | 19/63 | 16/61 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (any)=present at site of vaccination
Redness (mild) (Skin and subcutaneous tissue disorders) | 23/70 | 19/75 | 0/0 | 0/0 | 9/51 | 10/54 — Infant Series Dose 1 and Toddler Dose; Redness (mild)=0.5 to 2.0 cm
Redness (mild) (Skin and subcutaneous tissue disorders) | 18/61 | 24/65 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (mild)=0.5 to 2.0 cm
Redness (mild) (Skin and subcutaneous tissue disorders) | 12/60 | 15/60 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (mild)=0.5 to 2.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 4/69 | 3/70 | 0/0 | 0/0 | 8/50 | 3/50 — Infant Series Dose 1 and Toddler Dose; Redness (moderate)=2.5 to 7.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 4/56 | 3/59 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (moderate)=2.5 to 7.0 cm
Redness (moderate) (Skin and subcutaneous tissue disorders) | 7/61 | 3/54 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (moderate)=2.5 to 7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/67 | 0/70 | 0/0 | 0/0 | 0/49 | 0/50 — Infant Series Dose 1 and Toddler Dose; Redness (severe) >7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/55 | 0/59 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Redness (severe) >7.0 cm
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/58 | 0/53 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Redness (severe) >7.0 cm
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 11/69 | 9/72 | 0/0 | 0/0 | 7/51 | 10/51 — Infant Series Dose 1 and Toddler Dose; Fever 38 degrees C but 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 6/55 | 8/61 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever 38 degrees C but 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 8/59 | 5/54 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever 38 degrees C but 39 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 0/67 | 0/70 | 0/0 | 0/0 | 1/50 | 0/49 — Infant Series Dose 1 and Toddler Dose; Fever > 39 degrees C but 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 0/55 | 0/58 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 39 degrees C but 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 0/58 | 1/51 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 39 degrees C but 40 degrees C
Fever > 40 degrees C (General disorders) | 0/67 | 0/70 | 0/0 | 0/0 | 0/49 | 0/49 — Infant Series Dose 1 and Toddler Dose; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 0/55 | 0/58 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 0/58 | 0/51 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 40 degrees C
Decreased appetite (General disorders) | 23/71 | 22/76 | 0/0 | 0/0 | 13/57 | 15/54 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 16/59 | 28/63 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 14/61 | 16/57 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 38/77 | 56/79 | 0/0 | 0/0 | 18/59 | 21/56 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 25/62 | 36/67 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 13/62 | 25/60 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 37/75 | 30/77 | 0/0 | 0/0 | 11/52 | 8/52 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 17/59 | 16/61 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 18/61 | 12/57 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 28/74 | 38/76 | 0/0 | 0/0 | 11/54 | 20/58 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 18/60 | 27/66 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 10/61 | 17/58 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.